CLINICAL TRIAL: NCT05098535
Title: Remembering Risk Using Visual Risk Display of MINS to Obtain Informed Consent to Undergo Elective Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Michael McMullen, Assistant Professor, Department of Anesthesiology and Perioperative Medicine, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ANAE35219
Record Dates: First submitted 2021-07-29; First posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Risk
Keywords: Preoperative Assessment; Myocardial Injury; Perioperative Medicine; Personalized Medicine; Communication
MeSH Terms: conditions — Communication | interventions — Audiovisual Aids

STUDY DESIGN:
Intervention Model Description: A block randomized approach will be used to generate 2 groups of patients who will have their preoperative risk discussion guided by the use of a structured script or have the risk discussion guided by the use of a structured script and the display of a visual aid outlining the risk of myocardial injury.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be masked to the primary purpose of the study during their preoperative consultation. Upon receiving and completing the survey responses participants will be asked to recall their individualized risk of myocardial injury and provide feedback on the risk discussion they had with the anesthesiologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visual Aid + Scripted Risk Discussion (Experimental): This will involve the group of patients randomized to receive their perioperative risk discussion supplemented with the use of a visual aid in addition to a scripted discussion of their personalized perioperative risk of myocardial injury (MINS) during their consultation with an anesthesiologist in the PSS clinic.
  Interventions: Other: Visual Aid; Other: Scripted Risk Discussion
- Scripted Risk Discussion (Active Comparator): This will involve a group of patients randomized to receive a scripted discussion of their personalized perioperative risk of myocardial injury (MINS) during their consultation with an anesthesiologist in the PSS clinic.
  Interventions: Other: Scripted Risk Discussion

INTERVENTIONS:
Other: Visual Aid — The visual aid will include a graphic display of 100 individuals with number of individuals anticipated to suffer a myocardial injury highlighted by being filled in in red. There will also be a textual description stating the anticipated risk.
  For example in a patient with an rCRI score = 2 the text will state 10 out of 100 patients will have a myocardial injury (MINS) and 90 out of 100 patients will have no myocardial injury and 10 of the patients will be shaded red on the visual aid. The patients in this intervention will also received the scripted discussion of perioperative risk of MINS.
  Arms: Visual Aid + Scripted Risk Discussion
Other: Scripted Risk Discussion — The patients seen in PSS will have a standardized discussion of perioperative risk of myocardial injury read to them by the anesthesiologist in the PSS clinic.

SUMMARY:
Disclosure of anticipated risks to individuals considering undergoing an elective operative procedure is an important aspect of informed consent process. Recent Canadian Guidelines have highlighted the importance of perioperative risk discussion within the context of preoperative assessment but there is little prior research into potential interventions to optimize the communication of risks.

Myocaridal injury (MINS) is the most common complication and this study is focused on determining the effectiveness of current communication strategies in our presurgical consultations and to quantifying the impact of introducing a visual aid and scripted risk discussions has on patients ability to recall their individualized perioperative risk of myocardial injury.

DETAILED DESCRIPTION:
Informed consent is an important aspect of the patient-physician relationship. Prior to agreeing to undergo treatment patients must have risks and benefits disclosed to a "reasonable patient" standard.1 The 2016 Canadian Cardiovascular Society Guidelines on Perioperative Cardiac Risk Assessment made strong recommendations emphasizing the need for clear communication of perioperative cardiac risk to patients.2 Myocardial injury is the most common post-operative complications and has significant impact on patient outcomes including survival.2. However, very few studies have examined the communication of risk to patients, particularly when communicating perioperative cardiac risk.

The aim of this study is to formally evaluate the effectiveness of perioperative risk communication and examine if the introduction of visual aids can improve communication and preoperative patient education. During this study, all patients presenting to the Presurgical Screening clinic for consultation with an anesthesiologist will receive a standardized scripted discussion of the risk of myocardial injury following noncardiac surgery (MINS) based on their revised cardiac risk index. During the study period, patients will be randomized in blocks to exposure to a visual aid representing their individualized risk of MINS during the risk discussion. Immediately following the anesthesiology consultation, all patient will be invited to participate in the study and complete a survey that will assess ability to recall individualized cardiac risk and examine current risk discussion practices, patient satisfaction with cardiac risk discussion, importance of cardiac risk disclosure, assess anxiety related to risk discussion, and seek general feedback from participants. This study is structured to assess the effectiveness of incorporating the use of structured, scripted risk discussion with and without the use of a visual aid. A subset of consenting patients will be followed-up post operatively (within 48h) to assess recall of preoperative cardiac risk discussion.

The investigators hypothesizes that the use of visual representation of perioperative risk of Myocardial Injury after Non-Cardiac Surgery during the pre-anesthetic assessment will improve the patients' satisfaction with the cardiac risk discussion and the participant's understanding and retention of the risk in the post-operative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients 45 years of age or older
* Patient is assessed in person by an anesthesiologist at Presurgical Screening Clinic
* Patient schedule for elective non-cardiac surgery

Exclusion Criteria:

* Unable to provide consent due to communication/language barrier
* Prior enrollment in this study
* Unable to consent without a Substitute Decision Maker
* Scheduled for non-elective surgery

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-10-28 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Immediate Recall of Perioperative Risk of Myocardial Injury (MINS) | Within one hour of completing consultation with anesthesiologist in PSS clinic
  This will be calculated as the patients who can state their risk estimate within the 95% CI for the risk estimate given their rCRI score (as outlined in the 2016 CCS Guidelines) when completing the survey This will be calculated as the patients who can state their risk estimate within the 95% CI for the risk estimate given their rCRI score (as outlined in the 2016 CCS Guidelines) when completing the survey.

SECONDARY OUTCOMES:
Postoperative Recall of Perioperative Risk of Myocardial Injury (MINS) | Within 72h of undergoing their elective surgical procedure
  This will be calculated as the patients who can state their risk estimate within the 95% CI for the risk estimate given the participant's rCRI score (as outlined in the 2016 CCS Guidelines) when completing the survey
Demographics and Immediate Recall of Perioperative Risk of Myocardial Injury | Within one hour of completing preoperative consultation
  Investigators will compare the impact sex, age and level of education have on the percentage of patients able to recall their risk estimate within the 95% CI outlined in CCS guidelines
Correlation between subjective rating of individual risk and numeric risk estimate | Within one hour completing preoperative consultation
  Patients subjective responses to the level of risk (minimal, low, moderate, high, very high) will be compared with their numeric risk estimate ( rate / 100 persons)
Satisfaction with Risk Discussion | Within one hour completing preoperative consultation
  Subjects will be asked to rate the level of satisfaction with the preoperative risk discussion on a 5 point likehert scale and the difference between two groups will be examined
Recommendation of Use of Risk Discussion Tool in Future | Within one hour completing preoperative consultation
  Patients will be asked to rate the likelihood the participant would recommend (0-10) the use of a similar format of risk discussion to family or friends coming for surgery

CONTACTS AND LOCATIONS:
Overall Officials: Michael McMullen, MD, Principal Investigator — Queens University
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duceppe E, Parlow J, MacDonald P, Lyons K, McMullen M, Srinathan S, Graham M, Tandon V, Styles K, Bessissow A, Sessler DI, Bryson G, Devereaux PJ. Canadian Cardiovascular Society Guidelines on Perioperative Cardiac Risk Assessment and Management for Patients Who Undergo Noncardiac Surgery. Can J Cardiol. 2017 Jan;33(1):17-32. doi: 10.1016/j.cjca.2016.09.008. Epub 2016 Oct 4. PMID 27865641